CLINICAL TRIAL: NCT00668278
Title: I-Gel Versus Disposable Laryngeal Mask Airway for General Anesthesia With Controlled Ventilation
Brief Title: I-Gel Versus Disposable Laryngeal Mask (LMA) for General Anesthesia (GA) With Controlled Ventilation
Acronym: IGE(L)MA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Health and Social Care Trust (Other Government)
Collaborators: Antrim Area Hospital (Other)
Responsible Party: Dr William John Donaldson, Antrim Area Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 07/NIR01/124
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Healthy
Keywords: Supraglottic airway; I-gel; Laryngeal mask; Controlled ventilation; Peak airway pressure; Seal pressure; Anaesthesia; Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Laryngeal Mask Airway insertion
  Interventions: Device: Insertion of laryngeal mask airway (AuraOnce mask); Other: Measurement of airway pressures
- B (Active Comparator): I-gel insertion
  Interventions: Device: Insertion of I-gel airway; Other: Measurement of airway pressures

INTERVENTIONS:
Device: Insertion of laryngeal mask airway (AuraOnce mask) — Insertion of laryngeal mask airway under anaesthesia: Fentanyl 1-2mcg/kg; Propofol 1-3mg/kg; Atracurium 0.5mg/kg; AuraOnce disposable laryngeal mask
  Arms: A
Device: Insertion of I-gel airway — Insertion of I-gel airway under anaesthesia; Fentanyl 1-2mcg/kg; Propofol 1-3mg/kg; Atracurium 0.5mg/kg
  Arms: B
Other: Measurement of airway pressures — Measurement of peak airway pressure under steady state; measurement of device seal pressure

SUMMARY:
Randomized controlled trial comparing performance of the I-gel and disposable Laryngeal Mask Airways under controlled ventilation. 200 patients, 100 in each arm. Measurement of peak airway and sealing pressures. Postoperative questionnaires at 1 and 24hrs.

Hypothesis

There is no difference between the performance* of the I-gel and disposable laryngeal mask airways for controlled ventilation under general anesthesia.

*as defined by peak airway pressure and sealing pressures.

ELIGIBILITY:
Inclusion Criteria:

* Males and females.
* Age 18-89 inclusive.
* ASA grade 1-2.
* Elective surgery

Exclusion Criteria:

* Emergency surgery.
* Surgery within the peritoneum.
* Surgery requiring prone or steep head-down positioning.
* Patients at increased risk of aspiration

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Sealing pressure and peak airway pressure. | Under anaesthesia.

SECONDARY OUTCOMES:
Postoperative patient symptoms | 1hr and 24hrs postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: William J Donaldson, MBBS FRCA, Principal Investigator — Antrim Area Hospital, Northern Health and Social Care Trust, National Health Service, United Kingdom